CLINICAL TRIAL: NCT05355636
Title: The Effects of Fertility Management Counseling Supported With Telehealth on Contraceptive Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: contraceptive counseling
Record Dates: First submitted 2022-03-14; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-03

CONDITIONS: Counseling; Fertility; Contraception; Telehealth
Keywords: fertility management; counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (Experimental): patient receiving counseling
  Interventions: Behavioral: Fertility Management Counseling
- control group (No Intervention): patient without counseling

INTERVENTIONS:
Behavioral: Fertility Management Counseling — counseling
  Arms: experiment group

SUMMARY:
Fertility management refers to the entirety of practices that allow families to have as many children as they want and when they want, prevent unwanted pregnancies, regulate the time between two births and receive help in having children in the case of infertility.

According to the Turkey Demographic and Health Survey 2018 data, 70% of women in Turkey who are currently married do not use any contraceptive method. Based on the same data, the rate of the unmet need for fertility management is 12% nationwide, 14% in eastern provinces, and 17% in women at the ages of 20-24. These rates show that the rates of unmet fertility management needs in Turkey are still not on the desired level.

The fact that eastern provinces of Turkey have the lowest rate of modern contraceptive method use as 43% and a high rate of unmet fertility management needs as 14% suggests that it is needed to increase the effectiveness of fertility management counseling and reach more women. In these eastern provinces, especially women living in rural areas do not have easy access to these services due to the high prevalence of adolescent marriages, lack of transportation opportunities, healthcare personnel and healthcare services, and unpredictable weather conditions.

DETAILED DESCRIPTION:
To eliminate these obstacles to a relative extent, fertility management counseling will be provided through using the telehealth method. The World Health Organization states that telehealth practices will make access easier, eliminate geographical obstacles, increase the quality of healthcare, and allow the cost-effective management of the resources of the healthcare sector. The telehealth system increases the quality of healthcare, and thus, it has a significant role in managing the resources of the healthcare sector.

The Participant Information Form created by the researcher based on the review of the relevant literature includes questions about the sociodemographic characteristics of the participants (age, education level, employment status, income level) and pregnancy-related questions. The Contraceptive Method Usage Status Form (for the experimental and control groups) will be utilized to determine the contraceptive methods that are used by women in the 7th month of the postpartum period.The data that will be obtained in the study will be statistically analyzed using the International Business Machines Statistical Package for the Social Sciences Subscription Trial version. The analyses will include independent-samples t-test, ANOVA, and Cochran test. In cases of significant differences identified in ANOVA, Tukey's test will be used to identify the source of the difference in pairwise comparisons. The level of statistical significance is accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* volunteer
* be between the ages of 18-45
* to be primiparous
* have a smart phone
* complete education

Exclusion Criteria:

* refuse to research

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women between the ages of 18-45 who gave birth in primiparous
Enrollment: 70 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Telehealth on Contraceptive Use | 7 months
  The use of birth control methods by the fertility regulation consultancy service offered by Telehealth in postpartum women is a positive indicator of counseling.
Family Planning Method Using Status Form | 7 months
  It is a scale that examines the method use status of the participants after telehealth assisted fertility regulation counseling.

CONTACTS AND LOCATIONS:
Overall Officials: duygu tatar, MsC Student, Principal Investigator — Marmara University
Locations (1):
- Duygu Tatar, Bitlis, Bi̇tli̇s, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No